CLINICAL TRIAL: NCT04586049
Title: Autonomic Dysfunction, Brain Blood Flow and Cognitive Decline in Veterans With Gulf War Illness
Brief Title: Cardiovascular and Neurovascular Regulation in GWI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2019-0961; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); W81XWH1910381 (Other Grant/Funding Number: Department of Defense); Protocol Version 09/15/2021 (Other: UW Madison)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Brain Blood Flow; Neurovascular Control
Keywords: MRI; Brain Blood Flow; Sympathetic Nerve Activity; Cardiorespiratory Fitness
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Veterans with GWI: Veterans with GWI who served in the Gulf War between 1990 and 1992
  Interventions: Device: MRI; Device: Transcranial Doppler Ultrasound; Other: Sympathetic Nerve Activity
- Veterans without GWI (Controls): Veterans without GWI who served in the Gulf War between 1990 and 1992
  Interventions: Device: MRI; Device: Transcranial Doppler Ultrasound; Other: Sympathetic Nerve Activity

INTERVENTIONS:
Device: MRI — Participants will undergo an MRI scan while participating in a breathing test to measure brain blood flow.
Device: Transcranial Doppler Ultrasound — Participants will undergo a TCD scan while participating in a breathing test to measure brain blood flow.
Other: Sympathetic Nerve Activity — Participants will undergo sympathetic nerve activity testing while participating in a breathing test.

SUMMARY:
Brain blood flow regulation and autonomic dysfunction will be measured in Veterans with and without Gulf War Illness who served in the Gulf War between 1990 and 1992.

DETAILED DESCRIPTION:
Gulf War Illness (GWI) is a multi-symptom illness with unknown etiology. GWI is a leading cause of disability in Gulf War Veterans. Cognitive complaints are a common symptom of GWI, which suggests the brain is involved in the development of this condition. As Veterans age, these cognitive complaints may worsen and be compounded by the aging process. GWI may be a condition of "accelerated" brain aging. Therefore, there may be long-term consequences of GWI, and the presence of GWI may increase a person's risk for developing Alzheimer's Disease (AD) or other dementias. In comparison to other brain-related diseases such as stroke, relatively little is known about GWI and how this condition impacts the normal age-related changes in the brain.

The research aims are:

1. To determine if Veterans with Gulf War Illness demonstrate abnormal brain blood flow regulation and autonomic dysfunction when compared with Veterans without Gulf War Illness.
2. To determine if brain blood flow and autonomic nervous system variables in Veterans are associated with other markers of brain aging that are relevant to cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Deployed to the Persian Gulf between 1990-1992
* Body mass <300 lbs
* Diagnosis of Gulf War Illness based on CMI/CDC and Kansas definitions or No diagnosis of Gulf War Illness

Exclusion Criteria:

* Current or lifetime evidence of: Type II diabetes, neurological disease, cancer treatment, rheumatoid arthritis, lupus, bipolar disorder, psychotic disorders, or mood disorders with psychotic features
* Current illicit substance use or partial remission for less than 1 year
* Taking multiple sedatives or anticonvulsant medications
* Currently pregnant
* Absolute contraindications to exercise testing
* Contraindications to MRI
* Other significant medical conditions at investigator's discretion

Ages: 45 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will include Veterans with Gulf War Illness and Veterans without Gulf War Illness. Both men and women are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Brain blood flow measured using Transcranial Doppler ultrasound | Baseline
  Neurovascular control will be investigated by measuring the change in brain blood flow using a transcranial Doppler ultrasound in response to a breathing test.
Brain blood flow measured using MRI | Baseline
  Neurovascular control will be investigated by measuring the change in brain blood flow using an MRI in response to a breathing test.
Sympathetic nerve activity | Baseline
  Neurovascular control will be investigated by measuring the change in sympathetic nerve activity will be measured using microneurography in response to a breathing test.

CONTACTS AND LOCATIONS:
Overall Officials: Jill N Barnes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecrux C, Hamel E. The neurovascular unit in brain function and disease. Acta Physiol (Oxf). 2011 Sep;203(1):47-59. doi: 10.1111/j.1748-1716.2011.02256.x. Epub 2011 Mar 22. PMID 21272266
- [Background] Catchlove SJ, Parrish TB, Chen Y, Macpherson H, Hughes ME, Pipingas A. Regional Cerebrovascular Reactivity and Cognitive Performance in Healthy Aging. J Exp Neurosci. 2018 Jul 5;12:1179069518785151. doi: 10.1177/1179069518785151. eCollection 2018. PMID 30013388
- [Background] Lange G, Tiersky LA, Scharer JB, Policastro T, Fiedler N, Morgan TE, Natelson BH. Cognitive functioning in Gulf War Illness. J Clin Exp Neuropsychol. 2001 Apr;23(2):240-9. doi: 10.1076/jcen.23.2.240.1208. PMID 11309677
- [Background] Toomey R, Alpern R, Vasterling JJ, Baker DG, Reda DJ, Lyons MJ, Henderson WG, Kang HK, Eisen SA, Murphy FM. Neuropsychological functioning of U.S. Gulf War veterans 10 years after the war. J Int Neuropsychol Soc. 2009 Sep;15(5):717-29. doi: 10.1017/S1355617709990294. Epub 2009 Jul 29. PMID 19640317
- [Background] Bunegin L, Mitzel HC, Miller CS, Gelineau JF, Tolstykh GP. Cognitive performance and cerebrohemodynamics associated with the Persian Gulf Syndrome. Toxicol Ind Health. 2001 May;17(4):128-37. doi: 10.1191/0748233701th100oa. PMID 12479508
- [Background] Hubbard NA, Hutchison JL, Motes MA, Shokri-Kojori E, Bennett IJ, Brigante RM, Haley RW, Rypma B. Central Executive Dysfunction and Deferred Prefrontal Processing in Veterans with Gulf War Illness. Clin Psychol Sci. 2014 May 1;2(3):319-327. doi: 10.1177/2167702613506580. PMID 25767746
- [Background] Christova P, James LM, Engdahl BE, Lewis SM, Carpenter AF, Georgopoulos AP. Subcortical brain atrophy in Gulf War Illness. Exp Brain Res. 2017 Sep;235(9):2777-2786. doi: 10.1007/s00221-017-5010-8. Epub 2017 Jun 20. PMID 28634886
- [Background] Chao LL, Rothlind JC, Cardenas VA, Meyerhoff DJ, Weiner MW. Effects of low-level exposure to sarin and cyclosarin during the 1991 Gulf War on brain function and brain structure in US veterans. Neurotoxicology. 2010 Sep;31(5):493-501. doi: 10.1016/j.neuro.2010.05.006. Epub 2010 May 24. PMID 20580739
- [Background] Van Riper SM, Alexander AL, Koltyn KF, Stegner AJ, Ellingson LD, Destiche DJ, Dougherty RJ, Lindheimer JB, Cook DB. Cerebral white matter structure is disrupted in Gulf War Veterans with chronic musculoskeletal pain. Pain. 2017 Dec;158(12):2364-2375. doi: 10.1097/j.pain.0000000000001038. PMID 28796115
- [Background] Pop V, Sorensen DW, Kamper JE, Ajao DO, Murphy MP, Head E, Hartman RE, Badaut J. Early brain injury alters the blood-brain barrier phenotype in parallel with beta-amyloid and cognitive changes in adulthood. J Cereb Blood Flow Metab. 2013 Feb;33(2):205-14. doi: 10.1038/jcbfm.2012.154. Epub 2012 Nov 14. PMID 23149553
- [Background] Ikonomovic MD, Mi Z, Abrahamson EE. Disordered APP metabolism and neurovasculature in trauma and aging: Combined risks for chronic neurodegenerative disorders. Ageing Res Rev. 2017 Mar;34:51-63. doi: 10.1016/j.arr.2016.11.003. Epub 2016 Nov 6. PMID 27829172
- [Background] Johnson VE, Stewart W, Smith DH. Traumatic brain injury and amyloid-beta pathology: a link to Alzheimer's disease? Nat Rev Neurosci. 2010 May;11(5):361-70. doi: 10.1038/nrn2808. PMID 20216546
- [Background] Barnes JN. Exercise, cognitive function, and aging. Adv Physiol Educ. 2015 Jun;39(2):55-62. doi: 10.1152/advan.00101.2014. PMID 26031719
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Coverdale NS, Badrov MB, Shoemaker JK. Impact of age on cerebrovascular dilation versus reactivity to hypercapnia. J Cereb Blood Flow Metab. 2017 Jan;37(1):344-355. doi: 10.1177/0271678X15626156. Epub 2016 Jan 12. PMID 26759432
- [Background] Miller KB, Howery AJ, Harvey RE, Eldridge MW, Barnes JN. Cerebrovascular Reactivity and Central Arterial Stiffness in Habitually Exercising Healthy Adults. Front Physiol. 2018 Aug 17;9:1096. doi: 10.3389/fphys.2018.01096. eCollection 2018. PMID 30174609
- [Background] Barnes JN, Harvey RE, Miller KB, Jayachandran M, Malterer KR, Lahr BD, Bailey KR, Joyner MJ, Miller VM. Cerebrovascular Reactivity and Vascular Activation in Postmenopausal Women With Histories of Preeclampsia. Hypertension. 2018 Jan;71(1):110-117. doi: 10.1161/HYPERTENSIONAHA.117.10248. Epub 2017 Nov 20. PMID 29158356
- [Background] Kisler K, Nelson AR, Montagne A, Zlokovic BV. Cerebral blood flow regulation and neurovascular dysfunction in Alzheimer disease. Nat Rev Neurosci. 2017 Jul;18(7):419-434. doi: 10.1038/nrn.2017.48. Epub 2017 May 18. PMID 28515434
- [Background] Fabiani M, Gordon BA, Maclin EL, Pearson MA, Brumback-Peltz CR, Low KA, McAuley E, Sutton BP, Kramer AF, Gratton G. Neurovascular coupling in normal aging: a combined optical, ERP and fMRI study. Neuroimage. 2014 Jan 15;85 Pt 1(0 1):592-607. doi: 10.1016/j.neuroimage.2013.04.113. Epub 2013 May 9. PMID 23664952
- [Background] Girouard H, Iadecola C. Neurovascular coupling in the normal brain and in hypertension, stroke, and Alzheimer disease. J Appl Physiol (1985). 2006 Jan;100(1):328-35. doi: 10.1152/japplphysiol.00966.2005. PMID 16357086
- [Background] Janulewicz PA, Krengel MH, Maule A, White RF, Cirillo J, Sisson E, Heeren T, Sullivan K. Neuropsychological characteristics of Gulf War illness: A meta-analysis. PLoS One. 2017 May 17;12(5):e0177121. doi: 10.1371/journal.pone.0177121. eCollection 2017. PMID 28520755
- [Background] Haley RW, Spence JS, Carmack PS, Gunst RF, Schucany WR, Petty F, Devous MD Sr, Bonte FJ, Trivedi MH. Abnormal brain response to cholinergic challenge in chronic encephalopathy from the 1991 Gulf War. Psychiatry Res. 2009 Mar 31;171(3):207-20. doi: 10.1016/j.pscychresns.2008.05.004. Epub 2009 Feb 20. PMID 19230625
- [Background] Li X, Spence JS, Buhner DM, Hart J Jr, Cullum CM, Biggs MM, Hester AL, Odegard TN, Carmack PS, Briggs RW, Haley RW. Hippocampal dysfunction in Gulf War veterans: investigation with ASL perfusion MR imaging and physostigmine challenge. Radiology. 2011 Oct;261(1):218-25. doi: 10.1148/radiol.11101715. Epub 2011 Sep 13. PMID 21914840
- [Background] Liu P, Aslan S, Li X, Buhner DM, Spence JS, Briggs RW, Haley RW, Lu H. Perfusion deficit to cholinergic challenge in veterans with Gulf War Illness. Neurotoxicology. 2011 Mar;32(2):242-6. doi: 10.1016/j.neuro.2010.12.004. Epub 2010 Dec 13. PMID 21147163
- [Background] Falvo MJ, Lindheimer JB, Serrador JM. Dynamic cerebral autoregulation is impaired in Veterans with Gulf War Illness: A case-control study. PLoS One. 2018 Oct 15;13(10):e0205393. doi: 10.1371/journal.pone.0205393. eCollection 2018. PMID 30321200
- [Background] Joyner MJ, Casey DP. Regulation of increased blood flow (hyperemia) to muscles during exercise: a hierarchy of competing physiological needs. Physiol Rev. 2015 Apr;95(2):549-601. doi: 10.1152/physrev.00035.2013. PMID 25834232
- [Background] Barnes JN. Sex-specific factors regulating pressure and flow. Exp Physiol. 2017 Nov 1;102(11):1385-1392. doi: 10.1113/EP086531. Epub 2017 Sep 2. PMID 28799254
- [Background] Serrador JM, Picot PA, Rutt BK, Shoemaker JK, Bondar RL. MRI measures of middle cerebral artery diameter in conscious humans during simulated orthostasis. Stroke. 2000 Jul;31(7):1672-8. doi: 10.1161/01.str.31.7.1672. PMID 10884472
- [Background] Coverdale NS, Gati JS, Opalevych O, Perrotta A, Shoemaker JK. Cerebral blood flow velocity underestimates cerebral blood flow during modest hypercapnia and hypocapnia. J Appl Physiol (1985). 2014 Nov 15;117(10):1090-6. doi: 10.1152/japplphysiol.00285.2014. Epub 2014 Jul 10. PMID 25012027
- [Background] Berman SE, Rivera-Rivera LA, Clark LR, Racine AM, Keevil JG, Bratzke LC, Carlsson CM, Bendlin BB, Rowley HA, Blennow K, Zetterberg H, Asthana S, Turski P, Johnson SC, Wieben O. Intracranial Arterial 4D-Flow is Associated with Metrics of Brain Health and Alzheimer's Disease. Alzheimers Dement (Amst). 2015 Dec 1;1(4):420-428. doi: 10.1016/j.dadm.2015.09.005. PMID 26693176
- [Background] Rivera-Rivera LA, Turski P, Johnson KM, Hoffman C, Berman SE, Kilgas P, Rowley HA, Carlsson CM, Johnson SC, Wieben O. 4D flow MRI for intracranial hemodynamics assessment in Alzheimer's disease. J Cereb Blood Flow Metab. 2016 Oct;36(10):1718-1730. doi: 10.1177/0271678X15617171. Epub 2015 Nov 25. PMID 26661239
- [Background] White RF, Steele L, O'Callaghan JP, Sullivan K, Binns JH, Golomb BA, Bloom FE, Bunker JA, Crawford F, Graves JC, Hardie A, Klimas N, Knox M, Meggs WJ, Melling J, Philbert MA, Grashow R. Recent research on Gulf War illness and other health problems in veterans of the 1991 Gulf War: Effects of toxicant exposures during deployment. Cortex. 2016 Jan;74:449-75. doi: 10.1016/j.cortex.2015.08.022. Epub 2015 Sep 25. PMID 26493934
- [Background] Lucas KE, Armenian HK, Debusk K, Calkins HG, Rowe PC. Characterizing Gulf War Illnesses: neurally mediated hypotension and postural tachycardia syndrome. Am J Med. 2005 Dec;118(12):1421-7. doi: 10.1016/j.amjmed.2005.06.034. No abstract available. PMID 16378804
- [Background] Haley RW, Vongpatanasin W, Wolfe GI, Bryan WW, Armitage R, Hoffmann RF, Petty F, Callahan TS, Charuvastra E, Shell WE, Marshall WW, Victor RG. Blunted circadian variation in autonomic regulation of sinus node function in veterans with Gulf War syndrome. Am J Med. 2004 Oct 1;117(7):469-78. doi: 10.1016/j.amjmed.2004.03.041. PMID 15464703
- [Background] Peckerman A, LaManca JJ, Smith SL, Taylor A, Tiersky L, Pollet C, Korn LR, Hurwitz BE, Ottenweller JE, Natelson BH. Cardiovascular stress responses and their relation to symptoms in Gulf War veterans with fatiguing illness. Psychosom Med. 2000 Jul-Aug;62(4):509-16. doi: 10.1097/00006842-200007000-00009. PMID 10949096
- [Background] Peckerman A, Dahl K, Chemitiganti R, LaManca JJ, Ottenweller JE, Natelson BH. Effects of posttraumatic stress disorder on cardiovascular stress responses in Gulf War veterans with fatiguing illness. Auton Neurosci. 2003 Oct 31;108(1-2):63-72. doi: 10.1016/S1566-0702(03)00155-3. PMID 14614966
- [Background] Fukuda K, Nisenbaum R, Stewart G, Thompson WW, Robin L, Washko RM, Noah DL, Barrett DH, Randall B, Herwaldt BL, Mawle AC, Reeves WC. Chronic multisymptom illness affecting Air Force veterans of the Gulf War. JAMA. 1998 Sep 16;280(11):981-8. doi: 10.1001/jama.280.11.981. PMID 9749480
- [Background] Steele L. Prevalence and patterns of Gulf War illness in Kansas veterans: association of symptoms with characteristics of person, place, and time of military service. Am J Epidemiol. 2000 Nov 15;152(10):992-1002. doi: 10.1093/aje/152.10.992. PMID 11092441
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Cook DB, O'Connor PJ, Lange G, Steffener J. Functional neuroimaging correlates of mental fatigue induced by cognition among chronic fatigue syndrome patients and controls. Neuroimage. 2007 May 15;36(1):108-22. doi: 10.1016/j.neuroimage.2007.02.033. Epub 2007 Mar 3. PMID 17408973
- [Background] Staud R, Smitherman ML. Peripheral and central sensitization in fibromyalgia: pathogenetic role. Curr Pain Headache Rep. 2002 Aug;6(4):259-66. doi: 10.1007/s11916-002-0046-1. PMID 12095460
- [Background] Schweinhardt P, Bushnell MC. Pain imaging in health and disease--how far have we come? J Clin Invest. 2010 Nov;120(11):3788-97. doi: 10.1172/JCI43498. Epub 2010 Nov 1. PMID 21041961
- [Background] Barnes JN, Hart EC, Curry TB, Nicholson WT, Eisenach JH, Wallin BG, Charkoudian N, Joyner MJ. Aging enhances autonomic support of blood pressure in women. Hypertension. 2014 Feb;63(2):303-8. doi: 10.1161/HYPERTENSIONAHA.113.02393. Epub 2013 Dec 9. PMID 24324040
- [Background] Joyner MJ, Wallin BG, Charkoudian N. Sex differences and blood pressure regulation in humans. Exp Physiol. 2016 Mar;101(3):349-55. doi: 10.1113/EP085146. Epub 2015 Aug 16. PMID 26152788
- [Background] Barnes JN, Harvey RE, Eisenmann NA, Miller KB, Johnson MC, Kruse SM, Lahr BD, Joyner MJ, Miller VM. Cerebrovascular reactivity after cessation of menopausal hormone treatment. Climacteric. 2019 Apr;22(2):182-189. doi: 10.1080/13697137.2018.1538340. Epub 2019 Jan 21. PMID 30661405
- [Background] MacLeod CM. Half a century of research on the Stroop effect: an integrative review. Psychol Bull. 1991 Mar;109(2):163-203. doi: 10.1037/0033-2909.109.2.163. No abstract available. PMID 2034749
- [Background] Lucas SJ, Ainslie PN, Murrell CJ, Thomas KN, Franz EA, Cotter JD. Effect of age on exercise-induced alterations in cognitive executive function: relationship to cerebral perfusion. Exp Gerontol. 2012 Aug;47(8):541-51. doi: 10.1016/j.exger.2011.12.002. Epub 2012 Jan 2. PMID 22230488
- [Background] McMillan KM, Laird AR, Witt ST, Meyerand ME. Self-paced working memory: validation of verbal variations of the n-back paradigm. Brain Res. 2007 Mar 30;1139:133-42. doi: 10.1016/j.brainres.2006.12.058. Epub 2006 Dec 23. PMID 17280644
- [Background] Jaeggi SM, Schmid C, Buschkuehl M, Perrig WJ. Differential age effects in load-dependent memory processing. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2009;16(1):80-102. doi: 10.1080/13825580802233426. Epub 2008 Aug 5. PMID 18686052
- [Background] Rickards CA, Johnson BD, Harvey RE, Convertino VA, Joyner MJ, Barnes JN. Cerebral blood velocity regulation during progressive blood loss compared with lower body negative pressure in humans. J Appl Physiol (1985). 2015 Sep 15;119(6):677-85. doi: 10.1152/japplphysiol.00127.2015. Epub 2015 Jul 2. PMID 26139213
- [Background] Committee on Gulf War and Health: Treatment for Chronic Multisymptom Illness; Board on the Health of Select Populations; Institute of Medicine. Gulf War and Health: Treatment for Chronic Multisymptom Illness. Washington (DC): National Academies Press (US); 2013 Apr 4. Available from http://www.ncbi.nlm.nih.gov/books/NBK206744/ PMID 24901196